CLINICAL TRIAL: NCT02008344
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Favipiravir in Adult Subjects With Uncomplicated Influenza
Brief Title: Phase 3 Efficacy and Safety Study of Favipiravir for Treatment of Uncomplicated Influenza in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MDVI, LLC (Industry)
Collaborators: MediVector, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T705US317; U1111-1147-8470 (Other: UTN)
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: influenza; flu; fever; cough; body aches; headache; nasal congestion; body pains; sore throat; fatigue; T-705; favipiravir; favor; flu symptoms
MeSH Terms: conditions — Influenza, Human; Fever; Cough; Headache; Nasal Obstruction; Pharyngitis; Fatigue | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- favipiravir (Active Comparator): Day 1: 1800 mg (1st loading dose), 1800 mg (2nd loading dose) Days 2-5: 800 mg BID (3rd to 10th dose)
  Interventions: Drug: favipiravir
- placebo (Placebo Comparator): Day 1: 1800 mg (1st loading dose), 1800 mg (2nd loading dose) Days 2-5: 800 mg BID (3rd to 10th dose)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: favipiravir — Administered twice daily over 5 consecutive days for a total of 10 doses.
  * Day 1: 1800 mg twice daily (loading doses)
  * Days 2 through 5: 800 mg twice daily
  Other Names: T-705
  Arms: favipiravir
Drug: placebo — Administered twice daily over 5 consecutive days for a total of 10 doses.
  * Day 1: 1800 mg twice daily (loading doses)
  * Days 2 through 5: 800 mg twice daily
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if favipiravir is effective in reducing the time to resolution of influenza symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a 5-day regimen of favipiravir reduces the time to alleviation of influenza symptoms, resolution of fever, and viral shedding, in subjects with uncomplicated influenza compared to no treatment (e.g. placebo).

ELIGIBILITY:
Inclusion Criteria:

* At time of enrollment has 2 or more of the following symptoms (moderate to severe in intensity) that began 48 hours or less prior to the anticipated start of dosing with study medication: cough, sore throat, headache, nasal congestion, body aches and pains, fatigue
* Has a fever at the first visit or in the 6 hours prior if antipyretics were taken, defined as: ≥ 38.0°C (≥ 100.4°F) if < 65 years old; or ≥ 37.8°C (≥ 100.0°F) if ≥ 65 years old
* Tests positive for influenza A or B during the 48 hours between onset of symptoms and anticipated dosing with study medication as confirmed by RAT or PCR testing (study or non-study procedure); or per Investigator and Medical Monitor discretion in the event there is a known influenza outbreak circulating in the community or the subject has been in close contact with a person who was recently confirmed to have laboratory-confirmed influenza
* Willing to adhere to strict contraceptive measures throughout study and for 3 months following last dose of study medication

Exclusion Criteria:

* Female subjects who are pregnant, currently breast-feeding, or have a positive pregnancy test at Screening
* Has taken an anti-influenza drug, or received any live attenuated influenza vaccine within 4 weeks prior to signing the informed consent
* Has underlying chronic respiratory disease; includes bronchial asthma if currently experience asthma symptoms, requires current asthma treatment, or has had an asthma attack in the past year
* Is suspected of having bacterial respiratory infection (i.e., expectoration of purulent or mucopurulent sputum and/or infiltrate in lung observed on chest x ray, or is on antibiotics for pulmonary disease) at start of study
* Has a history of gout or is under treatment for: gout or hyperuricemia; hereditary xanthinuria; hypouricemia or xanthine calculi of the urinary tract
* Has a history of hypersensitivity to an anti-viral nucleoside-analog drug targeting a viral RNA polymerase
* Current use of adrenocorticosteroids (except topical preparation) or immunosuppressive drugs
* Has an allergy or contraindication to use of acetaminophen (paracetamol)
* Has a serious chronic disease, history of alcohol or drug abuse within preceding 2 years, psychiatric illness not well controlled (not on stable regimen > 1 year), or is deemed by the Investigator to be ineligible for any reason
* Previously participated in a clinical trial of favipiravir (T-705)
* Has renal insufficiency requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of all primary influenza symptoms and fever | 21 days
  Time from the start of study treatment until alleviation of all primary influenza symptoms (i.e. cough, sore throat, headache, nasal congestion, body aches and pains, fatigue) and to resolution of fever

SECONDARY OUTCOMES:
Time to alleviation of each of the primary influenza symptoms and fever | 21 days
  Time from the start of study treatment until alleviation of each of the following influenza symptoms (cough, sore throat, headache, nasal congestion, body aches and pains, and fatigue) and to resolution of fever
To characterize the PK of favipiravir when used under clinical conditions | 21 days

OTHER OUTCOMES:
Changes in viral load | 15 days
  Changes in viral load as measured from nasopharyngeal swabs
Safety | 21 days
  Adverse events and clinical laboratory tests for systemic safety including hematology, clinical chemistry, and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Carol Epstein, MD, Study Director — MediVector, Inc.
Locations (202):
- United States (126):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Camp Verde, Arizona
  - Mesa, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Chula Vista, California
  - Fountain Valley, California
  - Fresno, California
  - Garden Grove, California
  - Gold River, California
  - Harbor City, California
  - La Mesa, California
  - Lomita, California
  - Los Angeles, California
  - Modesto, California
  - North Hollywood, California
  - Northridge, California
  - Oceanside, California
  - Paramount, California
  - Roseville, California
  - San Diego, California
  - San Gabriel, California
  - Stockton, California
  - Upland, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Glenwood Springs, Colorado
  - Waterbury, Connecticut
  - Celebration, Florida
  - Clearwater, Florida
  - Delray Beach, Florida
  - Edgewater, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Lauderdale Lakes, Florida
  - Lynn Haven, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Orange, Florida
  - Saint Cloud, Florida
  - South Miami, Florida
  - Summerfield, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - Norcross, Georgia
  - Oakwood, Georgia
  - Riverdale, Georgia
  - Snellville, Georgia
  - Idaho Falls, Idaho
  - Twin Falls, Idaho
  - Brownsburg, Indiana
  - Evansville, Indiana
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Opelousas, Louisiana
  - Columbia, Maryland
  - Towson, Maryland
  - Watertown, Massachusetts
  - Worcester, Massachusetts
  - Madison Heights, Michigan
  - Troy, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - Butte, Montana
  - Missoula, Montana
  - Bellevue, Nebraska
  - Las Vegas, Nevada
  - Lodi, New Jersey
  - New York, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Huntersville, North Carolina
  - Lexington, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Toledo, Ohio
  - Wadsworth, Ohio
  - Ashland, Oregon
  - Belle Vernon, Pennsylvania
  - Clairton, Pennsylvania
  - Indiana, Pennsylvania
  - Scottdale, Pennsylvania
  - Smithfield, Pennsylvania
  - Tyrone, Pennsylvania
  - Uniontown, Pennsylvania
  - Cumberland, Rhode Island
  - Greenville, South Carolina
  - Greer, South Carolina
  - Murrells Inlet, South Carolina
  - North Myrtle Beach, South Carolina
  - Rock Hill, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Franklin, Tennessee
  - Jackson, Tennessee
  - Smyrna, Tennessee
  - Allen, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - McKinney, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sealy, Texas
  - Sugar Land, Texas
  - Victoria, Texas
  - Draper, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Newport News, Virginia
  - Spokane, Washington
- Argentina (10):
  - La Palta, Buenos Aires
  - Buenos Aires, Ciudad Autónoma de BuenosAires
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - Santa Fe, Santa Fe Province
  - Buenos Aires
  - Mar del Plata
  - Ramos Mejía
  - San Miguel de Tucumán
  - Vicente López
- Brazil (9):
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Curitiba, Paraná
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Brasília
- Canada (22):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Cambridge, Ontario
  - Corunna, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Sarnia, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Drummondville, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - Victoriaville, Quebec
  - Saskatoon, Saskatchewan
- Colombia (5):
  - Medellín, Antioquia
  - Bogotá, Cundinamarca
  - Cali, Valle de Cauca
  - Cali, Valle del Cauca Department
  - Medellín
- Santo Domingo, National District, Dominican Republic
- El Salvador (2):
  - Santa Tecla, La Libertad Department
  - San Salvador, San Salvador Department
- Guatemala City, Departamento de Guatemala, Guatemala
- Mexico (16):
  - Chihuahua City, Chihuahua
  - León, Guanajanto
  - León, Guanajuato
  - Acapulco de Juárez, Guerrero
  - El Salto, Jalisco
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Distrito Federal, Mexico City
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
  - Xalapa, Veracruz
  - Cuautitlán Izcalli
  - Guanajanto
  - Mexico City
  - Tlalnepantla
- Peru (8):
  - Arequipa, Arequipa
  - Cusco, Departamento de Cusco
  - Ica, Ica
  - Trujillo, La Libertad
  - Lima, Lima Province
  - Miraflores, Lima region
  - Loreto, Loreto
  - Piura, Piura
- Puerto Rico (2):
  - Manatí
  - San Juan

REFERENCES:
- [Derived] Hayden FG, Lenk RP, Stonis L, Oldham-Creamer C, Kang LL, Epstein C. Favipiravir Treatment of Uncomplicated Influenza in Adults: Results of Two Phase 3, Randomized, Double-Blind, Placebo-Controlled Trials. J Infect Dis. 2022 Nov 11;226(10):1790-1799. doi: 10.1093/infdis/jiac135. PMID 35639525